CLINICAL TRIAL: NCT04241679
Title: Feasibility of Auditory Nerve Test System for Optimization of Simultaneous Translabyrinthine Vestibular Schwannoma Resection With Cochlear Implantation
Brief Title: Auditory Nerve Test System During Vestibular Schwannoma Resection
Acronym: ANTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Cameron Wick, Assistant Professor, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201910197; G190197 (Other: FDA - Investigational Device Exemption)
Record Dates: First submitted 2019-11-05; First posted 2020-01-27 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Vestibular Schwannoma; Acoustic Neuroma; Sensorineural Hearing Loss; Asymmetric Sensorineural Hearing Loss; Cochlear Nerve Damage; Cochlear Nerve Deafness; Skull Base Neoplasms; Auditory; Nerve
Keywords: Cochlear implant; Vestibular schwannoma; Acoustic Neuroma; Sensorineural hearing loss; Asymmetric sensorineural hearing loss; Single-sided deafness; Auditory nerve
MeSH Terms: conditions — Neuroma, Acoustic; Hearing Loss, Sensorineural; Vestibulocochlear Nerve Injuries; Retrocochlear Diseases; Skull Base Neoplasms; Vestibulocochlear Nerve Diseases

STUDY DESIGN:
Intervention Model Description: Single arm study of 10 patients with no serviceable hearing due to small or medium sized vestibular schwannomas undergoing translabyrinthine resection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention Group (Experimental): Patients undergoing a translabyrinthine approach for vestibular schwannoma resection will have the health of their auditory nerve monitored during tumor dissection. If the auditory nerve is visually confirmed to be intact, then concurrent cochlear implantation will be performed.
  Interventions: Device: Auditory Nerve Test System

INTERVENTIONS:
Device: Auditory Nerve Test System — The Auditory Nerve Test System provides an electrically-evoked signal from within the cochlea to facilitate intraoperative auditory nerve monitoring. The auditory nerve can be measured both at the root entry zone of the brainstem (eCNAP) and with scalp electrodes (eABR). Data on the health of the auditory nerve will be collected immediately prior to tumor dissection, during tumor dissection, and immediately after tumor dissection. The main purpose of this study is to determine feasibility of this novel intraoperative monitoring protocol.
  Secondarily, if the auditory nerve is visually confirmed to be intact following tumor resection then the patients will receive a cochlear implant during the same surgery.

SUMMARY:
The Auditory Nerve Test System (ANTS) is a novel device that stimulates the auditory nerve much like a cochlear implant. The purpose of this study is to demonstrate feasibility of the ANTS during translabyrinthine surgery for vestibular schwannoma resection. If the auditory nerve is kept intact, then the patients will also receive a cochlear implant at the same time potentially alleviating the morbidities caused by a vestibular schwannoma and asymmetric sensorineural hearing loss.

DETAILED DESCRIPTION:
Many patients diagnosed with a vestibular schwannoma (also called acoustic neuroma) eventually lose hearing in the afflicted ear. Improvements in magnetic resonance imaging (MRI) have led to tumors being diagnosed at smaller sizes, however, this has not changed the eventual demise in hearing for most patients. Hearing loss leads to tinnitus, poor sound localization, difficulty hearing in background noise, and imbalance all of which contribute to the decreased quality of life associated with a vestibular schwannoma diagnosis.

Some tumors may be resected while maintaining the integrity of the auditory nerve. When a patient has hearing, the health of the auditory nerve can be monitored during the surgery through auditory-evoked (sound) measurements. When a patient has already lost their hearing or the surgical approach sacrifices all residual hearing, then auditory-evoked measurements can no longer be used and there is no way to monitor the auditory nerve aside from visual inspection.

The Auditory Nerve Test System (ANTS) is a novel device designed to facilitate electrically-evoked auditory nerve monitoring. The ANTS is comprised of three parts: a test electrode, connector cable, and stimulator box. The test electrode functions like a mini-cochlear implant placed within the cochlea during a translabyrinthine surgery. During tumor resection the test electrode electrically stimulates the auditory nerve allowing surgeons to monitor electrophysiologic data on the health of the auditory nerve. The primary goal of this study is to assess the ANTS during translabyrinthine vestibular schwannoma resections.

If patient are able to maintain an intact auditory nerve following vestibular schwannoma resection then a cochlear implant will be placed during the same surgery. Secondary outcomes measures will investigate cochlear implant outcomes and patient quality of life following this procedure and over the first year of using their cochlear implant. These secondary outcomes will be measured at 3-months, 6-months, and 12-months following cochlear implant activation. The test will assess how well the cochlear implant is working, the cochlear implant's impact on sound localization and hearing in background noise, and finally various aspects relevant to the patient's quality of life (tinnitus, balance, hearing, and overall quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Vestibular schwannoma (sporadic or Neurofibromastosis Type-2)
* 12 years of age or older
* Tumor size < 2.5 cm
* Non-serviceable ipsilateral hearing
* No prior cochlear implant or auditory brainstem implant use
* No prior microsurgery or stereotactic radiation for this tumor
* Patient decision and medical clearance for a translabyrinthine approach for tumor resection
* Willingness to comply with research protocol
* Reasonable expectations of cochlear implant performance
* Auditory nerve integrity visually confirmed following tumor resection

Exclusion Criteria:

* Pathology/tumors other than a vestibular schwannoma
* Younger than 12 years of age
* Tumor size > 2.5 cm
* Serviceable hearing in the tumor ear
* Prior cochlear implant use in either the contralateral or ipsilateral ear
* Prior microsurgery or stereotactic radiation for this tumor
* Unwilling to comply with research protocol
* Auditory nerve integrity cannot be visually confirmed after tumor resection

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Auditory Nerve Electrophysiology | Intraoperative testing
  Reliability of electrically-evoked direct auditory nerve monitoring at the brainstem (eCNAP) and far-field auditory brainstem response (eABR). The auditory nerve signal will be monitored before, during, and after vestibular schwannoma resection. Elements like signal amplitude, latency, and preservation of eABR waveforms III and V will be measured.

SECONDARY OUTCOMES:
Cochlear Implant Speech Performance | 3-months and 12-months after cochlear implant activation
  Speech performance measured in the CI-only condition using CNC Words, AzBio Sentences in Quiet, and AzBio Sentences in +10 dB SNR.
Sound Localization | Initial cochlear implant activation, then repeated at 6-months and 12-months after activation.
  Using an audio booth that contains a sound arc, patients will be asked to identify where a sound is coming from in the implant-on and implant-off conditions. This ability to localize is measured with a root-mean-square (RMS) error rate.
Quality of Life Following Vestibular Schwannoma Resection | Pre-operative baseline, then 3-months and 12-months post-operative
  Diagnosis and treatment of vestibular schwannomas can impact multiple aspects of a patient's quality of life. Using patient-reported outcome measures these aspects will be measured throughout their treatment course. The specific questionnaires will be: Speech, Spatial and Qualities of Hearing (SSQ), Hearing Handicap Inventory for Adults (HHIA), Tinnitus Handicap Inventory (THI), Dizziness Handicap Inventory (DHI), Penn Acoustic Neuroma Quality of Life (PANQOL), Cochlear Implant Quality of Life (CIQOL).

CONTACTS AND LOCATIONS:
Overall Officials: Cameron C Wick, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No